CLINICAL TRIAL: NCT01719601
Title: A Post-Marketing Surveillance (PMS) Study on the Safety and Effectiveness of Immediate Release Tapentadol Hydrochloride Among Adult Filipino Patients With Moderate to Severe Acute Non-Cancer Pain
Brief Title: A Safety and Effectiveness Study of Immediate Release Tapentadol Hydrochloride Among Filipino Patients With Moderate to Severe Acute Non-Cancer Pain
Status: Withdrawn | Type: Observational
Why Stopped: The company decided to cancel this study in conformity with PH FDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100919; R331333PAI4008 (Other: Janssen Pharmaceutica); TAP-C-12-PH-001-V02 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Moderate to Severe Acute Non-Cancer Pain
Keywords: Moderate to severe acute non-cancer pain; Immediate release tapentadol hydrochloride; Tapentadol IR; Nucynta IR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immediate release tapentadol: Patients will be taking immediate release tapentadol hydrochloride as per the product insert approved in Philippines.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Immediate release tapentadol hydrochloride will be administered as per the recommended doses approved in Philippines. The recommended oral starting dose is 25 mg, 50 mg or 100 mg every 4 to 6 hours depending on the initial pain intensity and thereafter, the dose will be adjusted to maintain adequate analgesia with acceptable tolerability. The dosing regimen will be individualized according to the severity of pain being treated, the previous treatment experience, and the ability to monitor patients.
  Other Names: Nucynta IR

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of immediate release tapentadol hydrochloride for the relief of moderate to severe acute non-cancer pain among Filipino patients.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (study conducted at multiple sites), observational study (study in which the investigators/ physicians observe the patients and measure their outcomes). The study will enroll approximately 100 patients who will be taking immediate release tapentadol hydrochloride with a dosing regimen stipulated in the product insert. As this is an observational study, assessment of patients will be based on the accepted clinical practice in the Philippines. Patients will be monitored at baseline (Day 1) and throughout the 28-day treatment period of tapentadol IR (Day 7, Day 14 and Day 28) for effectiveness with the help of short form Brief Pain Inventory questionnaire. Safety evaluations will include assessment of adverse events, clinical laboratory tests, and co-morbid conditions. The total study will be conducted for 3 years and the duration of treatment will be for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Filipino patients with moderate to severe non-cancer pain with an onset of 12 weeks or less from the baseline visit Patient is experiencing either an acute exacerbation of non-cancer pain or pain that has progressed to the point with the duration of at least 7 days and in the prescribing physician's judgment requires treatment with a Schedule II opioid
* Medically stable on the basis of routine physical examination, medical history, and vital signs at the time of baseline visit

Exclusion Criteria:

* Refuse to protocol-defined use of effective contraception
* Pregnant and lactating women
* Patients with severe renal and hepatic impairment, and having or suspected paralytic ileus
* Patients with conditions where drugs with mu-opioid receptor agonist activity are contraindicated
* Patients with acute intoxication with alcohol, hypnotics, centrally acting analgesics, or psychotropic drugs or receiving other mu-opioid receptor agonist analgesics, general anesthetics, phenothiazines, other tranquilizers, and sedatives
* Patients who are receiving Monoamine oxidase (MAO) inhibitors or who have taken them within the last 14 days
* Patients with documented history of increased intracranial pressure, impaired consciousness, coma and seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino patients with moderate to severe acute non-cancer pain and who are on the approved product label of Immediate release tapentadol hydrochloride
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events and adverse drug reactions | From the date of first exposure of patient to the study medication until 30 days after the last dose of the study medication and at anytime the investigator deems it as necessary, as assessed for 3 years

SECONDARY OUTCOMES:
The short form Brief Pain Inventory (BPI) questionnaire scores | Baseline (Day 1), Day 7, Day 14 and Day 28
  The short form BPI allows patients to rate the severity of their pain on a scale of 0 (no pain) to 10 (pain as bad as you can imagine) and the degree to which their pain interferes with common dimensions of feeling and function (general activity, walking, work, mood, enjoyment of life, relations with others, and sleep) on a scale of 0 (no interference) to 10 (interferes completely).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica